CLINICAL TRIAL: NCT06073899
Title: Biopsychosocial Factors in Resistance Exercise in Individuals with Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 7
Record Dates: First submitted 2023-09-25; First posted 2023-10-10 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Knee Pain

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigator administering Pressure Pain Threshold will be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Quiet Rest (No Intervention): Participants will sit quietly for two minutes, three times. Pressure pain threshold will be measured between each two-minute interval.
- High Fatigue Exercise (Experimental): Participants will perform a leg extension exercise in a machine with weight equipment to 65% of their 1-repetition maximum. Participants will complete this exercise for three sets until they report the exercise is "hard" (8/10 on the OMNI perceived exertion scale).
  Interventions: Other: Leg Extension Exercise
- Low Fatigue Exercise (Active Comparator): Participants will perform a leg extension exercise in a machine with weight equipment to 65% of their 1-repetition maximum. Participants will complete this exercise for three sets until they report the exercise is "somewhat easy" (4/10 on the OMNI perceived exertion scale).
  Interventions: Other: Leg Extension Exercise

INTERVENTIONS:
Other: Leg Extension Exercise — Participants will perform a concentric quadriceps contraction into terminal knee extension with weight equivalent to 65% of a1-repetition maximum.
  Arms: High Fatigue Exercise; Low Fatigue Exercise

SUMMARY:
The purpose of this research is to examine changes in pain sensitivity during high fatigue exercise, low fatigue exercise, and no treatment in individuals who are currently experiencing knee pain. Dosing dynamic resistance exercise intensity based on fatigue level is a novel, clinically feasible method. Dynamic resistance exercise at a high intensity (75% 1 repetition maximum (RM)) produces significant hypoalgesia at local sites compared to no treatment; however, dosing intensity based on 1RM can be challenging to implement in the clinical setting. Fatiguing endurance tasks produce local and systemic reductions in pressure pain threshold with low intensity isometric exercise completed until failure resulting in the largest exercise induced hypoalgesia effects. Fatigue may be an important mediator in pain response to exercise.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing knee pain symptom intensity rated as 3/10 or higher in the past 24 hours

Exclusion Criteria:

* non-English speaking
* history of knee surgery or fracture within the past 6 months
* history of quadriceps tendon rupture
* history of a chronic pain condition, such as fibromyalgia
* systemic medical conditions that affect sensation, such as uncontrolled diabetes or neurological conditions
* blood clotting disorder, such as hemophilia
* known presence of cardiovascular, pulmonary, or metabolic disease
* current use of tobacco products
* contraindication to the application of ice, including blood pressure over 140/90 mmHg, -conditions that cause hives or blood in urine when exposed to cold, and any reductions in blood flow to arms or legs.
* not physically ready to exercise without a medical exam as indicated by the Physical Activity Readiness Questionnaire + (PAR-Q+)
* pain during active knee range of motion 0-90 degrees (examined during screening)
* Pregnant
* unable to attend 4 sessions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold | This procedure will be completed two times before and after each set of exercise with the average analyzed. Outcomes are examined during each intervention visit from enrollment to study completion, about 2 years.
  A computerized pressure algometer (AlgoMed, Ramat Yishai, Israel) with a 1 cm diameter rubber tip will be applied at a constant rate. Participants will be instructed to say 'stop' or 'pain' or press a response button connected to the algometer so that stimulus can be terminated when the sensation first changes from pressure to pain (pain threshold). This will be applied to the quadriceps and upper trapezius on the same side as the participant's knee pain.

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Wilson, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No